CLINICAL TRIAL: NCT04806724
Title: Opening the Conversation for Couples With Reproductive Health Concerns
Brief Title: Opening the Conversation Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Jessica Gorman, Associate Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 7621; HE-2022-41
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Program #1 (Experimental): Participants attend 5 sessions (1.5 hours each) consisting of education and skills training to address cancer-related reproductive and sexual health concerns. Sessions occur via videoconference.
  Interventions: Behavioral: Opening the Conversation
- Program #2 (Active Comparator): Participants attend 4 sessions (1.5 hours each) consisting of education and skills training to address cancer-related concerns. Sessions occur via videoconference.
  Interventions: Behavioral: Side by Side

INTERVENTIONS:
Behavioral: Opening the Conversation — The intervention includes 5 weekly sessions (1.5 hours each), plus participant educational materials, and is delivered to couples via videoconference by a trained interventionist. Participants are asked to complete home activities between sessions. Sessions focus on development of communication and coping skills, with a focus on reproductive and sexual health distress.
  Arms: Program #1
Behavioral: Side by Side — The intervention includes 4 weekly sessions (1.5 hours each), plus participant educational materials, and is delivered to couples via videoconference by a trained interventionist. Participants are asked to complete home activities between sessions. Sessions focus on development of communication and coping skills, with a focus on general cancer-related distress.
  Arms: Program #2

SUMMARY:
Young adult survivors of breast and gynecologic cancer face a number of challenges, including interrupted life plans. As many as two-thirds of these young survivors experience negative effects of cancer and cancer treatment on their reproductive health, including sexual function and ability to have children. These are among the most distressing aspects of life after cancer for young survivors and their partners, and when left unaddressed, lead to poorer mental health and quality of life. Yet, surprisingly, evidence-based programs are not available to help young couples manage this aspect of life after cancer. In this study, we will adapt and evaluate an intervention designed to help young couples cope with and communicate about cancer-related reproductive and sexual health concerns.

DETAILED DESCRIPTION:
The specific aims of the study are:

Aim 1 (Phase I). Systematically adapt an empirically supported couple-based skills training intervention to help young breast and gynecologic cancer (BGC) survivors and their partners jointly manage the reproductive and sexual health consequences of cancer.

Aim 2 (Phase II - Quantitative). Evaluate the efficacy of the intervention and hypothesized mediators by conducting a randomized trial. We will evaluate the efficacy of the newly adapted intervention, Opening the Conversation (OC), on survivors' and their partners' reproductive and sexual distress as well as the relationship, sexual, and psychosocial health outcomes. We will determine whether dyadic coping and communication mediate intervention effects on survivors' and partners' reproductive and sexual distress.

Aim 3 (Phase II - Qualitative). Evaluate couples' experiences within and across conditions to gain in-depth knowledge of intervention components that influence hypothesized mediators and outcomes.

ELIGIBILITY:
Inclusion Criteria:

Cancer survivor participants:

* Cancer diagnosis between ages 18-39 years
* Current age 18-44
* Cancer diagnosis 6 months-5 years prior to enrollment
* Diagnosed with breast and/or gynecologic cancer
* Cancer stage 1-4
* Ability to participate in a videoconference intervention
* Has committed partner willing to participate
* English speaking
* High speed internet access via smart phone, tablet and/or computer

Partner participants:

* Age 18 or older
* English speaking
* Ability to participate in a videoconference intervention
* High speed internet access via smart phone, tablet and/or computer

Exclusion Criteria:

-Cancer survivors and partners are excluded if either partner does not meet eligibility criteria. Both partners must enroll or the dyad will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in reproductive distress | Baseline to 3 months post-intervention
  Relationship concern domain of the Fertility Problem Inventory (FPI) scale. 10 items. Range 10-60. Higher score indicates more reproductive distress.
Change in sexual distress | Baseline to 3 months post-intervention
  Sexual and relationship distress (SaRDS). 30 items. Range 1-30. Higher score indicates more sexual distress.

SECONDARY OUTCOMES:
Change in relationship quality | Baseline to 3 months post-intervention
  Dyadic Adjustment Scale (DAS-7). 7 items. Range 0- 36. Higher score indicates higher relationship quality.
Change in relationship Intimacy | Baseline to 3 months post-intervention
  Miller Social Intimacy Scale (MSIS). 17 items. Range 17-170. Higher score indicates higher levels of intimacy.
Change in sexual function (female) | Baseline to 3 months post-intervention.
  Female Sexual Function Index (FSFI).19 items. Range 2-36. Higher score indicates higher functioning.
Chang in sexual function (male) | Baseline to 3 months post-intervention
  International Index of Erectile Function (IIEF). 15 items. Range 1-75. Higher score indicates a higher level of sexual functioning.
Change in global sexual satisfaction | Baseline to 3 months post-intervention
  Global Measure of Sexual Satisfaction (GMSEX). 5 items. Higher score indicates higher level of sexual satisfaction.
Change in depressive symptoms | Baseline to 3 months post-intervention
  Patient Health Questionnaire (PHQ-8).8 items. Range 0 -24. Higher score indicates higher levels of depression.
Change in global health-related quality of life | Baseline to 3 months post-intervention
  PROMIS Global 10 v1.2. Raw scores (range 10-50) are translated to T scores following PROMIS guidelines. Higher score indicates better functioning.
Change in self-efficacy to communicate about sex and intimacy (survivor only) | Baseline to 3 months post-intervention
  SECSI. 10 items. Range 0-30. Higher score indicates higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Gorman, PhD, MPH, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorman JR, Lyons KS, Harvey SM, Acquati C, Salsman JM, Kashy DA, Drizin JH, Smith E, Flexner LM, Hayes-Lattin B, Reese JB. Opening the Conversation: study protocol for a Phase III trial to evaluate a couple-based intervention to reduce reproductive and sexual distress among young adult breast and gynecologic cancer survivor couples. Trials. 2022 Sep 2;23(1):730. doi: 10.1186/s13063-022-06665-3. PMID 36056413